CLINICAL TRIAL: NCT04722913
Title: Cervicogenic Headache Among Subjects With Forward Head Posture: a Correlational Cross-sectional Study.
Brief Title: Relation Between Cervicogenic Headache and Forward Head Posture
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merna ibrahim, Researcher, Cairo University
Other Study IDs: CGH among subjects with FHP
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Photogrametry , flexion rotation (FRT) test, Diagnosis of CGH according diagnostic criteria of the Cervicogenic Headache International Study Group (CHISG) — Photogrammetry is the science and technology of obtaining reliable information about physical objects and the environment through the process of recording, measuring and interpreting photographic images and patterns of electromagnetic radiant imagery and other phenomena.
  Flexion rotation (FRT) test:
  FRT is a manual examination technique with high sensitivity and specificity. It is performed with the patient in supine by passively taking the cervical spine into full flexion. End-range cervical flexion imparts ligamentous tension that impedes movement at vertebral segments below C2.7 Maintaining the flexion position, the patient's head is then rotated to each side until the patient reports pain or the operator determines that end of motion has been achieved. It is then determined if a restriction in ROM is present.

SUMMARY:
This study will be designed to determining whether there is a relationship between CGH and cervical posture which may potentially provide physical therapists with evidence supporting the assessment and treatment of abnormal posture in this patient group.

DETAILED DESCRIPTION:
Headaches have been posed to be a common occurring complaint being as frequent as 66% in general population. One the common types of headaches is Cervicogenic Headache which is considered as a secondary headache whereas the symptoms occur due to cervical spine and its bony components, disc or soft tissue structures. Cervicogenic headache is a syndrome described as pain felt on one side of the head, relating same side neck, shoulder and arm pain that is aggravated by neck movements or sustained head posture The prevalence of CGH has been reported 4.1% in general population 17.5% in patients and 41.4% in medical students.

The most general cause of cervicogenic headache (CGH) is the alteration of structure in the neck due to bad posture.

Proper posture is defined as a musculoskeletal balance which involves a minimal amount of stress and strain on the body , Forward head posture (FHP) is one of the commonly recognized types of poor head postures in the sagittal plane.FHP was defined as 'any alignment in which the external auditory meatus is positioned anterior to the plumbline through the shoulder joint.

Sustaining the head in this forward posture for prolonged period of time has been associated with the development of other musculoskeletal disorders such as 'upper crossed syndrome', which leads to reduction of lordosis in lower cervical and kyphosis of upper thoracic vertebra. In the long run, this may cause shortening of muscular fibers muscles involving the atlanto-occipital articulation, overstretching of muscles around joint and leads to chronic neck pain , There are many factors that could contribute to the development of forward head posture such as age, gender frequency of physical activity, occupation, usage of computer and smartphones and others.

It is noted that CGHs can often be related to forward neck and head posture, which is accompanied by a high muscular tone of the supporting extensors to keep the head from gravity. Such unstable state causes overstrain of the cervical muscles, and induces headache and neck pain.

FHP is a common postural defect among university students. This high prevalence may be related to the prolonged computer use and faulty posture during lectures.

Office workers of being sedentary for prolonged periods are liable to adopt forward head posture and thus generating neck strain, sprain and pain. Moreover, forward head posture is commonly found in people spending long periods on computers, mobile phones and game consoles.

Cervical dysfunction from abnormal posture has been proposed to aggravate or cause CGH, but there are conflicting reports as to whether there is an association between posture and CGH.

Statement of the problem:

There is lack of literature concerning the presence of cervicogenic headache among subjects with forward head posture.

This study will answer the following question Does forward head Posture is associated with cervicogenic headache?

Purpose of the study:

This study will be designed to determining whether there is a relationship between CGH and cervical posture which may potentially provide physical therapists with evidence supporting the assessment and treatment of abnormal posture in this patient group.

Significance of the study:

Ideal posture describes a state of maintaining balance in the body using minimal musculoskeletal activity without causing pain or discomfort. The tendency to stay seated for long periods of time can cause changes in the alignment of the spine, leading to improper posture, such as a rounded shoulder or forward head posture (FHP) .This change in posture can lead to a spatial change between the spine and the line of gravity, causing an overload on muscles and connective tissues . Neck pain or neck dysfunction is a musculoskeletal disorder caused by improper posture with physical impairment or functional limitation. The FHP is known as an internal factor that causes dysfunction with shoulder and neck pain. FHP results in a posture in which the extended head and upper cervical, and the lower cervical vertebrae flex. This increases the length of the external moment (the arm) by moving the gravitational center (the head) ahead of the load bearing axis. The exposure to this constant load on the craniovertebral extension muscles and the noncontractile structures causes a change in the biomechanical movement, and this increased stress can cause musculoskeletal damage or pain. In addition, FHP can also limit the functional movement in the head and neck area. These limitations are caused by irregular rotation and gliding movement inside the articular capsule whilst moving the joint. Moreover, it was reported that extended periods of FHP can result in a decreased number of sarcomere, as well as shortening of the muscle fibers, which can affect muscular contraction. As mentioned above, there are frequent occurrences of functional movement limitations or non-specific pain in the head and neck region in patients with FHP. Therefore, many studies have described the aspects of FHP that lead to functional movement limitations, and the pain in the head and neck area.

It is known that the quality of life in people suffering from headache is worse than in healthy subjects, in addition, this high prevalence disorder has negative health consequences in terms of occupational, economic and social factors.

The proposed association between abnormal cervical posture and headache has been demonstrated in migraine and tension-type headaches, but there are conflicting results in CGH. Despite this lack of agreement, clinicians routinely assess and treat altered posture for CGH. therefore, it is important to examine possible associations in order to guide treatment.

Hypotheses:

There will be no significant relationship between cervicogenic headache and forward head posture.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Craniovertebral angle (CVA) less than 50 degrees. (Gavin Morrison, 2018).
2. University students who were taking consecutive lectures for 3 hours and who worked forward for 3 hours or more on laptop (Arfa Naz et al, 2018).

Exclusion Criteria:

1. History of signiﬁcant medical conditions that might be potential contraindications to physical examination of the cervical spine, including known cancer, osteoporosis, nerve root symptoms, inﬂammatory or infectious diseases affecting the neck instability of the cervical spine, or reported potential vertebrobasilar insufﬁciency symptoms (Peter K. Farmer et al, 2015).
2. History of cervical spine injures (fracture, sprain, strain, whiplash), cervical spondylosis, obvious spinal deformities, neurological and neuromuscular disorders, TMJ dysfunction, cervicothoracic and lumbar kyphoscoliosis, rheumatic disease, torticollis, and balance disorders (B. Shaghayegh fard et al, 2015).

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: University students who were taking consecutive lectures for 3 hours. Subjects who worked forward for 3 hours or more on laptop. Subjects usually in awkward head position.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
comparing FRT and photogrammetry findings to CHISG criteria. | baseline
  Analysis of photogrammetry, interpreting the results of the flexion rotation test to diagnose the presence of forward head posture then identify if FHP is correlated with cervicogenic headeach which will be diagnosed by diagnostic criteria of the Cervicogenic Headache International Study Group (CHISG).

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Ramzy, Professor, Study Director — Cairo University; Maher El-Kabalawy, Professor, Study Chair — Cairo University
Locations (1):
- Mirna Ebrahim Abdelmagid, Giza, Egypt

REFERENCES:
- [Background] Blumenfeld A, Siavoshi S. The Challenges of Cervicogenic Headache. Curr Pain Headache Rep. 2018 Jun 13;22(7):47. doi: 10.1007/s11916-018-0699-z. PMID 29900508